CLINICAL TRIAL: NCT03728868
Title: Tolerability and Risk of Adverse Events With a Probiotic Supplement: A Randomised and Placebo Controlled Study in Healthy Individuals
Brief Title: Tolerability and Risk of Adverse Events With a Probiotic Supplement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: MetaboGen AB (Industry)
Responsible Party: Principal Investigator, Mattias Lorentzon, Professor, Chief physician, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: META002
Record Dates: First submitted 2018-10-02; First posted 2018-11-02 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Healthy Individuals
Keywords: Faecalibacterium prausnitzii; Desulfovibrio piger; tolerability; blood glucose levels

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): One capsule containing placebo (identical to the capsule with active product (F. prausnitzii and D. piger) in taste and appearance but without the active component) taken orally once a day (morning), one hour before breakfast on empty stomach, for 8 consecutive weeks.
  Interventions: Dietary Supplement: Placebo
- High dose F. prausnitzii and D. piger (Active Comparator): One capsule (containing F. prausnitzii and D. piger at a dose of 1E9-5x1E9 colony forming units per bacterial strain) taken orally once a day (morning), one hour before breakfast on empty stomach, for 8 consecutive weeks.
  Interventions: Dietary Supplement: High dose F. prausnitzii and D. piger
- Low dose F. prausnitzii and D. piger (Active Comparator): One capsule (containing F. prausnitzii and D. piger at a dose of 1E8-5x1E8 colony forming units per bacterial strain) taken orally once a day (morning), one hour before breakfast on empty stomach, for 8 consecutive weeks.
  Interventions: Dietary Supplement: Low dose F. prausnitzii and D. piger

INTERVENTIONS:
Dietary Supplement: Placebo — Dietary supplementation with placebo once a day for 8 consecutive weeks
  Arms: Placebo
Dietary Supplement: High dose F. prausnitzii and D. piger — Dietary supplementation with high dose F. prausnitzii and D. piger once a day for 8 consecutive weeks
  Arms: High dose F. prausnitzii and D. piger
Dietary Supplement: Low dose F. prausnitzii and D. piger — Dietary supplementation with low dose F. prausnitzii and D. piger once a day for 8 consecutive weeks
  Arms: Low dose F. prausnitzii and D. piger

SUMMARY:
The butyrate-producing bacterium Faecalibacterium prausnitzii is abundant in the human bowel and can make up to 5% of the gastrointestinal flora in healthy individuals. A reduced presence of it has been associated with an imbalance in the gastrointestinal flora of metabolic syndromes such as type 2 diabetes, fat liver, and in inflammatory bowel disease.

The present double-blind, placebo-controlled, randomized study is designed to investigate if dietary supplementation with F.prausnitzii (combined with D. piger) once a day for 8 consecutive weeks is tolerated compared to placebo and if it can affect the metabolism in a positive way.

DETAILED DESCRIPTION:
The understanding of the role of the gastrointestinal microbes for human health has gained considerable interest in recent years. The butyrate-producing bacterium Faecalibacterium prausnitzii is a naturally occurring bacterial species in the human gut that can make up to 5% of the gastrointestinal flora in healthy individuals.

Several studies have shown that the presence of butyrate producing bacteria, including F. prausnitzii, is lower in patients with inflammatory bowel disease; Crohn's disease and ulcerative colitis. Furthermore, lower levels of short fatty acids have been found in people with ulcerative colitis as compared to healthy individuals. Similar results have been obtained from studies about Crohn's disease, where people with a low abundance of F. prausnitzii run a higher risk of post-operative recurrence of their disease.

It has become evident that bacteria in the human gastrointestinal tract are symbiotic and dependent on each other's metabolism. Studies conducted by the sponsor (Metabogen AB) have shown that butyrate production from F. prausnitzii increases in the presence of Desulfovibrio piger, a common sulphate-reducing bacterium present in the human intestine. The symbiotic relationship between F. prausnitzii and D. piger can be utilised by combining these bacterial species into a probiotic dietary supplement, thus maintaining butyrate production in the intestine.

In animal models, who received approximately 5,000 times higher doses per kilogram of body weight than the highest dose scheduled in the proposed study, the intake of F. prausnitzii has shown anti-inflammatory effects as well as positive effects on the metabolism.

The present study is a double-blind, placebo-controlled, randomized, study in 48 healthy individuals (men and women) between 20 and 40 years old recruited from the general population. These volunteers will either receive F. prausnitzii and D. piger (in two different doses) or placebo orally once a day for 8 consecutive weeks. The investigators will assess how well treatment with the study product compared to placebo is tolerated (termination due to adverse events within 8 weeks of treatment) and if it can cause gastrointestinal symptoms (measured with The Gastrointestinal Symptom Rating Scale). The investigators will also assess if the intake of the study product can potentially give positive effects in the metabolism (blood glucose, fatty acids, protein ect).

ELIGIBILITY:
Inclusion Criteria:

1. 20 to 40 years old
2. Signed consent for participation
3. Healthy individuals without any known diseases
4. Willingness and ability to attend to planned visits, participate in telephone interviews and follow study instructions
5. Understanding the Swedish language in spoken and written terms

Exclusion Criteria:

1. Ongoing treatment with prescription drugs
2. Regular or sporadic intake of probiotic products (foods with probiotics are allowed)
3. Treated with antibiotics during the last 3 months
4. Pregnancy
5. Have experienced gastrointestinal tract symptoms (during the last month), which could affect study participation, as deemed by study physician.
6. Current tobacco use (smoking or snuff)
7. Participation in another clinical study

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Tolerability of the oral intake of F. prausnitzii and D. piger, defined as study discontinuation due to adverse events under 8 weeks of treatment. | 0-8 weeks
  How well treatment with the study product compared to placebo is tolerated, which is primarily defined as termination due to adverse events under 8 weeks of treatment.

SECONDARY OUTCOMES:
Gastrointestinal side effects, measured using the Gastrointestinal Symptom Rating Scale (GSRS) | 0-8 weeks
  Gastrointestinal symptoms are measured with The Gastrointestinal Symptom Rating Scale (GSRS), which includes 15 items combined into five symptom clusters measuring 1) reflux, 2) abdominal pain, 3) indigestion, 4) diarrhoea and 5) constipation. GSRS has a seven-point graded Likert-type scale, in which 1 represents absence of troublesome symptoms and 7 represents very troublesome symptoms. The total score is derived from all subclasses, resulting in a score between 0 and 45.
Effects on inflammation - erythrocyte sedimentation rate (safety parameters ) | 0-8 weeks
  Change in erythrocyte sedimentation rate in blood. Significant change in erythrocyte sedimentation rate before and after the 8-week treatment period.
Effects on inflammation - CRP (safety parameters ) | 0-8 weeks
  Change in C-reactive protein (CRP) level in blood. Significant change in CRP before and after the 8-week treatment period.
Effect on hematopoiesis - red blood cells (safety parameters) | 0-8 weeks
  Changes in red blood cells count. Significant change in red blood cell count before and after the 8-week treatment period.
Effect on hematopoiesis - white blood cells (safety parameters) | 0-8 weeks
  Changes in white blood cells count. Significant change in white blood cells count before and after the 8-week treatment period.
Effect on hematopoiesis - platelets (safety parameters) | 0-8 weeks
  Changes in platelets count. Significant change in platelets count before and after the 8-week treatment period.
Effects on liver enzymes - ALAT (safety parameters) | 0-8 weeks
  Changes in liver enzyme ALAT (Alanine transaminase). Significant changes before baseline and after 8 weeks of treatment.
Effects on liver enzymes - ASAT (safety parameters) | 0-8 weeks
  Changes in liver enzyme ASAT (Aspartate transaminase). Significant changes before baseline and after 8 weeks of treatment.
Effects on liver enzymes - ALP (safety parameters) | 0-8 weeks
  Changes in liver enzyme, ALP (Alkaline phosphatase). Significant changes before baseline and after 8 weeks of treatment.
Effects on serum bilirubin (safety parameters) | 0-8 weeks
  Changes in serum bilirubin. Significant changes before baseline and after 8 weeks of treatment.
Effects on the blood glucose | 0-8 weeks
  Changes (in percent) in levels of fasting blood glucose and HbA1c before and after the 8 week treatment period.
Effects on abundance of short-chain fatty acids | 0-10 weeks
  Changes in short-chain fatty acids in stool from baseline to week 10.
Colonization with F. prausnitzii | 0-8 weeks
  Colonization of the intestine with the total amount of F. prausnitzii bacteria. Measured in stool.
Effect on renal function(safety parameter) | 0-8 weeks
  Change in calculated eGFR (Glomerular Filtration Rate, based on serum creatinine)
Effect on serum total protein (safety parameter) | 0-8 weeks
  Change in serum total protein

CONTACTS AND LOCATIONS:
Overall Officials: Mattias Lorenzon, MD, PhD, Principal Investigator — Dept Geriatrics, Sahlgrenska University Hospital
Locations (1):
- Geriatric Medicine, Sahlgrenska University Hospital, Mölndal, Gothenburg, Västra Götaland County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Backhed F, Ding H, Wang T, Hooper LV, Koh GY, Nagy A, Semenkovich CF, Gordon JI. The gut microbiota as an environmental factor that regulates fat storage. Proc Natl Acad Sci U S A. 2004 Nov 2;101(44):15718-23. doi: 10.1073/pnas.0407076101. Epub 2004 Oct 25. PMID 15505215
- [Background] Turnbaugh PJ, Hamady M, Yatsunenko T, Cantarel BL, Duncan A, Ley RE, Sogin ML, Jones WJ, Roe BA, Affourtit JP, Egholm M, Henrissat B, Heath AC, Knight R, Gordon JI. A core gut microbiome in obese and lean twins. Nature. 2009 Jan 22;457(7228):480-4. doi: 10.1038/nature07540. Epub 2008 Nov 30. PMID 19043404
- [Background] Smith MI, Yatsunenko T, Manary MJ, Trehan I, Mkakosya R, Cheng J, Kau AL, Rich SS, Concannon P, Mychaleckyj JC, Liu J, Houpt E, Li JV, Holmes E, Nicholson J, Knights D, Ursell LK, Knight R, Gordon JI. Gut microbiomes of Malawian twin pairs discordant for kwashiorkor. Science. 2013 Feb 1;339(6119):548-54. doi: 10.1126/science.1229000. Epub 2013 Jan 30. PMID 23363771
- [Background] Le Chatelier E, Nielsen T, Qin J, Prifti E, Hildebrand F, Falony G, Almeida M, Arumugam M, Batto JM, Kennedy S, Leonard P, Li J, Burgdorf K, Grarup N, Jorgensen T, Brandslund I, Nielsen HB, Juncker AS, Bertalan M, Levenez F, Pons N, Rasmussen S, Sunagawa S, Tap J, Tims S, Zoetendal EG, Brunak S, Clement K, Dore J, Kleerebezem M, Kristiansen K, Renault P, Sicheritz-Ponten T, de Vos WM, Zucker JD, Raes J, Hansen T; MetaHIT consortium; Bork P, Wang J, Ehrlich SD, Pedersen O. Richness of human gut microbiome correlates with metabolic markers. Nature. 2013 Aug 29;500(7464):541-6. doi: 10.1038/nature12506. PMID 23985870
- [Background] Karlsson FH, Tremaroli V, Nookaew I, Bergstrom G, Behre CJ, Fagerberg B, Nielsen J, Backhed F. Gut metagenome in European women with normal, impaired and diabetic glucose control. Nature. 2013 Jun 6;498(7452):99-103. doi: 10.1038/nature12198. Epub 2013 May 29. PMID 23719380
- [Background] Qin J, Li Y, Cai Z, Li S, Zhu J, Zhang F, Liang S, Zhang W, Guan Y, Shen D, Peng Y, Zhang D, Jie Z, Wu W, Qin Y, Xue W, Li J, Han L, Lu D, Wu P, Dai Y, Sun X, Li Z, Tang A, Zhong S, Li X, Chen W, Xu R, Wang M, Feng Q, Gong M, Yu J, Zhang Y, Zhang M, Hansen T, Sanchez G, Raes J, Falony G, Okuda S, Almeida M, LeChatelier E, Renault P, Pons N, Batto JM, Zhang Z, Chen H, Yang R, Zheng W, Li S, Yang H, Wang J, Ehrlich SD, Nielsen R, Pedersen O, Kristiansen K, Wang J. A metagenome-wide association study of gut microbiota in type 2 diabetes. Nature. 2012 Oct 4;490(7418):55-60. doi: 10.1038/nature11450. Epub 2012 Sep 26. PMID 23023125
- [Background] Ott SJ, Musfeldt M, Wenderoth DF, Hampe J, Brant O, Folsch UR, Timmis KN, Schreiber S. Reduction in diversity of the colonic mucosa associated bacterial microflora in patients with active inflammatory bowel disease. Gut. 2004 May;53(5):685-93. doi: 10.1136/gut.2003.025403. PMID 15082587
- [Background] Loomba R, Seguritan V, Li W, Long T, Klitgord N, Bhatt A, Dulai PS, Caussy C, Bettencourt R, Highlander SK, Jones MB, Sirlin CB, Schnabl B, Brinkac L, Schork N, Chen CH, Brenner DA, Biggs W, Yooseph S, Venter JC, Nelson KE. Gut Microbiome-Based Metagenomic Signature for Non-invasive Detection of Advanced Fibrosis in Human Nonalcoholic Fatty Liver Disease. Cell Metab. 2017 May 2;25(5):1054-1062.e5. doi: 10.1016/j.cmet.2017.04.001. PMID 28467925
- [Background] Hsiao EY, McBride SW, Hsien S, Sharon G, Hyde ER, McCue T, Codelli JA, Chow J, Reisman SE, Petrosino JF, Patterson PH, Mazmanian SK. Microbiota modulate behavioral and physiological abnormalities associated with neurodevelopmental disorders. Cell. 2013 Dec 19;155(7):1451-63. doi: 10.1016/j.cell.2013.11.024. Epub 2013 Dec 5. PMID 24315484
- [Background] Machiels K, Joossens M, Sabino J, De Preter V, Arijs I, Eeckhaut V, Ballet V, Claes K, Van Immerseel F, Verbeke K, Ferrante M, Verhaegen J, Rutgeerts P, Vermeire S. A decrease of the butyrate-producing species Roseburia hominis and Faecalibacterium prausnitzii defines dysbiosis in patients with ulcerative colitis. Gut. 2014 Aug;63(8):1275-83. doi: 10.1136/gutjnl-2013-304833. Epub 2013 Sep 10. PMID 24021287
- [Background] Sokol H, Pigneur B, Watterlot L, Lakhdari O, Bermudez-Humaran LG, Gratadoux JJ, Blugeon S, Bridonneau C, Furet JP, Corthier G, Grangette C, Vasquez N, Pochart P, Trugnan G, Thomas G, Blottiere HM, Dore J, Marteau P, Seksik P, Langella P. Faecalibacterium prausnitzii is an anti-inflammatory commensal bacterium identified by gut microbiota analysis of Crohn disease patients. Proc Natl Acad Sci U S A. 2008 Oct 28;105(43):16731-6. doi: 10.1073/pnas.0804812105. Epub 2008 Oct 20. PMID 18936492
- [Derived] Khan MT, Dwibedi C, Sundh D, Pradhan M, Kraft JD, Caesar R, Tremaroli V, Lorentzon M, Backhed F. Synergy and oxygen adaptation for development of next-generation probiotics. Nature. 2023 Aug;620(7973):381-385. doi: 10.1038/s41586-023-06378-w. Epub 2023 Aug 2. PMID 37532933